CLINICAL TRIAL: NCT05040841
Title: Supporting Sustained HIV Treatment Adherence After Initiation
Acronym: SUSTAIN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Desmond Tutu HIV Foundation (Other); Massachusetts General Hospital (Other); New York University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: H-41920; 1R01MH125703-01A1 (NIH)
Record Dates: First submitted 2021-09-01; First posted 2021-09-10 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: HIV Infections; Adherence, Medication
Keywords: HIV treatment; HIV treatment adherence; Retention in care; Randomized controlled trial; Fractional factorial design; Proctor implementation science framework; Cost-effectiveness; South Africa; Community clinics
MeSH Terms: conditions — HIV Infections; Medication Adherence

STUDY DESIGN:
Intervention Model Description: The investigators will randomize subjects to one of 16 conditions, using a fractional factorial design to determine the effects of five intervention components.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Condition 1 (Experimental): Includes 1 intervention:
  S2/Peer: Enhanced peer group support.
  Interventions: Behavioral: S2/Peer: Enhanced peer group support
- Condition 2 (Experimental): Includes 1 intervention:
  S1/Text: Weekly check-in text messages.
  Interventions: Behavioral: S1/Text: Weekly check-in texts
- Condition 3 (Experimental): Includes 1 intervention:
  M3/EAM: Electronic adherence monitoring (EAM) + outreach to the patient.
  Interventions: Behavioral: M3/EAM: Immediate outreach to subject after EAM-identified missed doses
- Condition 4 (Experimental): Includes 3 interventions:
  M3/EAM: Electronic adherence monitoring (EAM) + outreach to the patient; S1/Text: Weekly check-in text messages; S2/Peer: Enhanced peer group support.
  Interventions: Behavioral: M3/EAM: Immediate outreach to subject after EAM-identified missed doses; Behavioral: S1/Text: Weekly check-in texts; Behavioral: S2/Peer: Enhanced peer group support
- Condition 5 (Experimental): Includes 1 intervention:
  M2/PRM: Pharmacy refill monitoring (PRM) + outreach to the patient.
  Interventions: Behavioral: M2/PRM: Immediate outreach to subject after a missed pharmacy refill
- Condition 6 (Experimental): Includes 3 interventions:
  M2/PRM: Pharmacy refill monitoring (PRM) + outreach to the patient S1/Text: Weekly check-in text messages; S2/Peer: Enhanced peer group support.
  Interventions: Behavioral: M2/PRM: Immediate outreach to subject after a missed pharmacy refill; Behavioral: S1/Text: Weekly check-in texts; Behavioral: S2/Peer: Enhanced peer group support
- Condition 7 (Experimental): Includes 3 interventions:
  M2/PRM: Pharmacy refill monitoring (PRM) + outreach to the patient M3/EAM: Electronic adherence monitoring (EAM) + outreach to the patient; S2/Peer: Enhanced peer group support.
  Interventions: Behavioral: M2/PRM: Immediate outreach to subject after a missed pharmacy refill; Behavioral: M3/EAM: Immediate outreach to subject after EAM-identified missed doses; Behavioral: S2/Peer: Enhanced peer group support
- Condition 8 (Experimental): Includes 3 interventions:
  M2/PRM: Pharmacy refill monitoring (PRM) + outreach to the patient; M3/EAM: Electronic adherence monitoring (EAM) + outreach to the patient; S1/Text: Weekly check-in text messages.
  Interventions: Behavioral: M2/PRM: Immediate outreach to subject after a missed pharmacy refill; Behavioral: M3/EAM: Immediate outreach to subject after EAM-identified missed doses; Behavioral: S1/Text: Weekly check-in texts
- Condition 9 (Experimental): Includes 1 intervention:
  M1/OTR: Outreach (OTR) to patient due to unsuppressed VL test result.
  Interventions: Behavioral: M1/OTR: Immediate outreach to subject due to unsuppressed viral load test result
- Condition 10 (Experimental): Includes 3 interventions:
  M1/OTR: Outreach to patient due to unsuppressed VL test result; S1/Text: Weekly check-in text messages; S2/Peer: Enhanced peer group support.
  Interventions: Behavioral: M1/OTR: Immediate outreach to subject due to unsuppressed viral load test result; Behavioral: S1/Text: Weekly check-in texts; Behavioral: S2/Peer: Enhanced peer group support
- Condition 11 (Experimental): Includes 3 interventions:
  M1/OTR: Outreach to patient due to unsuppressed VL test result; M3/EAM: Electronic adherence monitoring (EAM) + outreach to the patient; S2/Peer: Enhanced peer group support.
  Interventions: Behavioral: M1/OTR: Immediate outreach to subject due to unsuppressed viral load test result; Behavioral: M3/EAM: Immediate outreach to subject after EAM-identified missed doses; Behavioral: S2/Peer: Enhanced peer group support
- Condition 12 (Experimental): Includes 3 interventions:
  M1/OTR: Outreach to patient due to unsuppressed VL test result; M3/EAM: Electronic adherence monitoring (EAM) + outreach to the patient; S1/Text: Weekly check-in text messages.
  Interventions: Behavioral: M1/OTR: Immediate outreach to subject due to unsuppressed viral load test result; Behavioral: M3/EAM: Immediate outreach to subject after EAM-identified missed doses; Behavioral: S1/Text: Weekly check-in texts
- Condition 13 (Experimental): Includes 3 interventions:
  M1/OTR: Outreach to patient due to unsuppressed VL test result; M2/PRM: Pharmacy refill monitoring (PRM) + outreach to the patient; S2/Peer: Enhanced peer group support.
  Interventions: Behavioral: M1/OTR: Immediate outreach to subject due to unsuppressed viral load test result; Behavioral: M2/PRM: Immediate outreach to subject after a missed pharmacy refill; Behavioral: S2/Peer: Enhanced peer group support
- Condition 14 (Experimental): Includes 3 interventions:
  M1/OTR: Outreach to patient due to unsuppressed VL test result; M2/PRM: Pharmacy refill monitoring (PRM) + outreach to the patient; S1/Text: Weekly check-in text messages.
  Interventions: Behavioral: M1/OTR: Immediate outreach to subject due to unsuppressed viral load test result; Behavioral: M2/PRM: Immediate outreach to subject after a missed pharmacy refill; Behavioral: S1/Text: Weekly check-in texts
- Condition 15 (Experimental): Includes 3 interventions:
  M1/OTR: Outreach to patient due to unsuppressed VL test result; M2/PRM: Pharmacy refill monitoring (PRM) + outreach to the patient; M3/EAM: Electronic adherence monitoring (EAM) + outreach to the patient.
  Interventions: Behavioral: M1/OTR: Immediate outreach to subject due to unsuppressed viral load test result; Behavioral: M2/PRM: Immediate outreach to subject after a missed pharmacy refill; Behavioral: M3/EAM: Immediate outreach to subject after EAM-identified missed doses
- Condition 16 (Experimental): Includes 5 interventions:
  M1/OTR: Outreach to patient due to unsuppressed VL test result; M2/PRM: Pharmacy refill monitoring (PRM) + outreach to the patient; M3/EAM: Electronic adherence monitoring (EAM) + outreach to the patient; S1/Text: Weekly check-in text messages; S2/Peer: Enhanced peer group support.
  Interventions: Behavioral: M1/OTR: Immediate outreach to subject due to unsuppressed viral load test result; Behavioral: M2/PRM: Immediate outreach to subject after a missed pharmacy refill; Behavioral: M3/EAM: Immediate outreach to subject after EAM-identified missed doses; Behavioral: S1/Text: Weekly check-in texts; Behavioral: S2/Peer: Enhanced peer group support

INTERVENTIONS:
Behavioral: M1/OTR: Immediate outreach to subject due to unsuppressed viral load test result — Standard of care viral loads are drawn at month 4, month 12 and annually thereafter. Those with a raised viral load are often not immediately recalled, but identified at their next visit (1-2 months later) and asked to attend the "Risk of Treatment Failure" (ROTF) clinic for adherence support when they next attend. For subjects assigned to M1 we will add a call or other outreach (e.g., text, Whatsapp, in accordance with the outreach methods subjects indicate are appropriate for them at the Enrollment visit); to the subject as soon as a raised viral load result is received (±3-5 days), thus expediting entry to existing adherence support. There are two chances to be identified as nonadherent and linked immediately to existing adherence support in the first 12 months of care with M1.
  Other Names: M1/OTR
  Arms: Condition 10; Condition 11; Condition 12; Condition 13; Condition 14; Condition 15; Condition 16; Condition 9
Behavioral: M2/PRM: Immediate outreach to subject after a missed pharmacy refill — The subject will be contacted if he/she fails to collect medication from the pharmacy. A subject who is ≥7 days late for a monthly medication pick-up or 14 days late for a 2-monthly pick-up will be notified, again expediting entry to existing adherence support. There are 8-10 chances of being identified as nonadherent and linked immediately to existing adherence support in the first 12 months of care with M2.
  Other Names: M2/PRM
  Arms: Condition 13; Condition 14; Condition 15; Condition 16; Condition 5; Condition 6; Condition 7; Condition 8
Behavioral: M3/EAM: Immediate outreach to subject after EAM-identified missed doses — The subject will be contacted if he/she misses ≥4 doses or any three consecutive doses in a 14-day period, reviewed weekly, as identified by the EAM (electronic adherence monitor). There are 52 chances of being identified as nonadherent and linked immediately to existing adherence support in the first 12 months of care with M2.
  Other Names: M3/EAM
  Arms: Condition 11; Condition 12; Condition 15; Condition 16; Condition 3; Condition 4; Condition 7; Condition 8
Behavioral: S1/Text: Weekly check-in texts — Subject will receive weekly check-in texts in addition to the core adherence support component in the event they are identified as nonadherent and are linked with the Risk of Treatment Failure clinics. Subjects will be sent weekly simple but supportive text messages e.g. "how are you?" with the offer of a follow-up voice call for 16 consecutive weeks after being identified as nonadherent.
  Other Names: S1/Text
  Arms: Condition 10; Condition 12; Condition 14; Condition 16; Condition 2; Condition 4; Condition 6; Condition 8
Behavioral: S2/Peer: Enhanced peer group support — Subject will receive an enhanced form of peer group support. Standard of care Basic peer groups are led by lay counsellors and provide social support and education; this will continue to be provided to all patients who are not assigned to the enhanced version. "Enhanced" peer group support will replace the Basic standard of care 4 x 60 minute peer groups; and aim to improve long-term maintenance of adherence through motivational interviewing over 4-8 weeks.
  Other Names: S2/Peer
  Arms: Condition 1; Condition 10; Condition 11; Condition 13; Condition 16; Condition 4; Condition 6; Condition 7

SUMMARY:
The investigators will implement a 24-month fractional factorial design study (Aim 1). The investigators will recruit 510 patients initiating antiretroviral therapy (ART) at three City of Cape Town ART clinics. Each patient will have adherence monitored using the Wisepill® electronic adherence monitoring device (EAM). After eligibility has been confirmed, each participant will be randomized to one of 16 experimental conditions. Each condition includes a unique combination of five adherence intervention components. Three of these components focus on identifying individuals with poor adherence, with increasing degrees of sophistication, with immediate linkage to adherence support. Two components focus on supporting good adherence. They both supplement the existing adherence support program delivered at the study clinics operated by City of Cape Town (standard of care component). Based on Self-Determination Theory, the investigators postulate these intervention components will: 1) enhance feelings of autonomy support, social support, and knowledge; 2) improve motivation and self-competence; and 3) increase ART retention, adherence, and viral suppression. A subset of the participants, as well as clinic staff, will be invited to in-depth interviews to explore mediating factors (Aim 1) and the implementation process (Aim 2); and the data collected in Aims 1 and 2 will be used to explore cost effectiveness (Aim 3).

DETAILED DESCRIPTION:
The study's primary research goal is to identify the optimal combination of evidence-based and scalable HIV interventions for low-resource, high-burden settings. The investigators propose to 1) test the relative contribution of five promising intervention components; 2) collect cost and other implementation data; and 3) create a multi-component intervention package to optimize cost-effectiveness and implementation success. Of the five components, three are methods of non-adherence detection plus patient outreach; two are adherence support methods that can be integrated into Cape Town healthcare systems. These will not overcome all challenges that ART patients experience (e.g., structural barriers such as food insecurity) but they represent scalable, feasible, acceptable, and effective options. Notably, they are all behavioral approaches grounded in the experience and priorities of local health officials with whom the investigators have worked to identify scaleable interventions. While the study will be in Cape Town, it is broadly adaptable to other resource-limited settings.

The gold standard for testing interventions is the randomized controlled trial (RCT), which minimizes bias when testing cause and effect of a new exposure. When testing an intervention with more than one element, however, untangling the effect of individual elements is impossible. Indeed, data on the performance of individual components and their interactions-critical for developing and refining the components of a packaged intervention-is lost in an RCT. Notably, clinical care typically relies on packages of services, not single interventions, and packaged interventions are recommended for ART support. An effective way to test a multi-component intervention is to use the novel Multiphase Optimization STrategy (MOST), an engineering-inspired method for identifying the most efficacious combination of components in a packaged intervention, thus allowing researchers to drop inactive or weakly-performing components and construct an optimized package based on effect, cost, and other features. Once the optimized multi-component intervention is chosen, an RCT or quasi-experiment can follow to determine whether the optimized package yields superior outcomes compared to existing standards. MOST encompasses three phases: 1) preparation; 2) optimization; and 3) evaluation, often in an RCT. In this project, we have completed preparation, including a pilot study in Cape Town. SUSTAIN will comprise the middle optimization phase. The evaluation phase will be the focus of a future study.

The specific aims are:

Aim 1. Employ a highly efficient fractional factorial design to determine the effects of five intervention components on the primary outcome (HIV viral suppression) and secondary outcomes (ART adherence measured by EAM, ART retention per clinic records, days of unsuppressed virus, time to nonadherence detection, and time to linkage to support). The investigators will explore effect mechanisms quantitatively and qualitatively.

Aim 2. Evaluate the intervention components to address implementation, service, and client outcomes according to the Proctor framework. Data collection will involve tracking of intervention component use, time and motion studies, and quantitative surveys and qualitative interviews with participants and staff.

Aim 3. Use the effectiveness data collected in Aim 1 and the implementation and client outcomes in Aim 2 to model the multi-component intervention optimized for cost-effectiveness and implementation success.

Study Summary This study is designed to advance the translation of evidence-based interventions into clinical settings to benefit patients. There is ample evidence on what works to support ART adherence and retention-much of it from our own research. The investigators partnered with local officials and clinical staff in Cape Town to review the evidence and to conduct formative research to identify the most effective, acceptable, and feasible intervention options for patients and providers. The proposed study represents the next critical step: the investigators will test the intervention components that emerged from the formative work, encompassing elements to both rapidly identify nonadherent patients and to strengthen the support they receive once identified, to provide the data needed to construct the most cost-effective and sustainable multi-component intervention. The choice of intervention components will allow a critical test of advanced monitoring technology compared to simpler tools to identify nonadherence. By using an innovative MOST design to guide collection and analysis of efficacy, cost, and other implementation data, the study aligns with NIH's goals of using novel scientific methods to advance implementation science.

ELIGIBILITY:
Inclusion Criteria - Main study:

* Adults (≥18 years) and adolescents 16-17 years.
* HIV-positive and attending a local City of Cape Town (COCT) clinic to commence ART.
* Able to provide full informed consent, with a written signature. For those who are illiterate, a witness will be present throughout the process and will sign the form, while the participant will add their right thumb print. For those who are aged 16-17 years, informed written assent will be obtained, and the adolescent must have a parent or guardian who can provide full informed consent (see **below for how parent/guardian is defined for this purpose).
* Access to a working cellphone and willingness to receive study-related messaging on that phone.
* Willingness to comply with study procedures, including providing regular updates of contact details /locator information, and use a EAM device for the duration of participation.

Other Inclusion Criteria:

Aim 1: In-depth interviews (IDIs) with subset of trial subjects at baseline and months 12 and 24.

* Participation in the main trial.
* Self-reported prior experience with substance use, depression, gender inequity, stigma, or transport/clinic issues.

Aim 2: Questionnaires and IDIs with staff members at study clinics (three total clinics).

* Adults (≥18 years)
* Staff at study clinics, providing HIV care and/or treatment.

Aim 2: Focus group discussion (FGD) with City of Cape Town officials.

* Adults (≥18 years)
* Staff at City of Cape Town.

Exclusion Criteria - Main study:

* Clinical conditions as assessed by the COCT clinic clinicians at first visit e.g. renal disease, which preclude the use of a single tablet regimen (with the exception of those on tuberculosis (TB) treatment who are required to take an extra dose of dolutegravir daily).
* Planning to leave Cape Town permanently within the next 24 months.
* Being perinatally infected with HIV. Being infected from birth typically means a set of experiences and complications at a young age that require unique and special attention.
* If an adolescent, taking their ART medication as a syrup, as they are required to use the electronic adherence monitor (Wisepill device), which is only suitable for tablets.

Other Inclusion Criteria:

Aim 1: IDIs with trial subjects.

• None.

Aim 2: Questionnaires and IDIs with staff members at clinics. • None.

Aim 2: FGD with City of Cape Town officials.

• None.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
HIV viral suppression at 24 months | 24 months
  This outcome will measure the effect of the interventions on HIV viral suppression from enrollment to the end of study participation. HIV viral suppression will be defined as % plasma viral load (VL) <50 copies/mL (dichotomous).

SECONDARY OUTCOMES:
HIV viral suppression at 12 months | 12 months
  This outcome will be an intermediary outcome measure performed half-way through study participation. HIV viral suppression will be defined as % plasma VL <50 copies/mL (dichotomous).
Change in HIV viral load between baseline and 12 months | baseline, 12 months
  This will measure the effect on HIV viral load of exposure to interventions during the first half of study participation. It will be measured as the change in HIV viral load, defined as the mean change in HIV plasma between month 0 and month 12 post-enrollment (continuous).
Change in HIV viral load between baseline and 24 months | baseline, 24 months
  This will measure the effect on HIV viral load of exposure to interventions over the entire course of study participation. It will be measured as the change in HIV viral load, defined as the mean change in HIV plasma between month 0 and month 24 post-enrollment (continuous).
Days of unsuppressed virus between baseline and 24 months | baseline, 24 months
  This measure will determine the days that subjects experience unsuppressed virus, measured between baseline and the end of the study at 24 months (continuous).
Achievement of ≥ 90% adherence in month 24 | month 24
  This measure indicates whether subject achieved adherence of 90% or more during the final month of study participation in month 24 (dichotomous).
Mean adherence from baseline through 24 months | baseline through 24 months
  This measure indicates mean adherence over the entire length of the study from enrollment through 24 months (continuous).

CONTACTS AND LOCATIONS:
Overall Officials: Lora Sabin, PhD, MA, Principal Investigator — Boston University
Locations (3):
- South Africa (3):
  - Mzamomhle, Cape Town, Western Cape
  - Phumlani, Cape Town, Western Cape
  - Weltevreden Valley, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: No
We have not yet made a detailed plan, but tentatively, we will deposit de-identified IPD in a repository at Boston University (BU) School of Public Health and the Desmond Tutu Health Foundation that can be made available to other researchers once our planned analyses are complete.

REFERENCES:
- [Derived] Jennings L, West RL, Halim N, Kaiser JL, Gwadz M, MacLeod WB, Gifford AL, Haberer JE, Orrell C, Sabin LL. Protocol for an evaluation of adherence monitoring and support interventions among people initiating antiretroviral therapy in Cape Town, South Africa-a multiphase optimization strategy (MOST) approach using a fractional factorial design. Trials. 2023 May 5;24(1):310. doi: 10.1186/s13063-023-07322-z. PMID 37147725